CLINICAL TRIAL: NCT06372366
Title: Oral Manifestations in a Group of Egyptian Children With Short Stature and a Group of Healthy Egyptian Children : A Cross Sectional Study
Brief Title: Oral Manifestations in Egyptian Children With Short Stature
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Soliman Abd El-Ghaffar Abd El-Megid Abd Allah, Principal researcher (Dentist), Cairo University
Other Study IDs: Oral signs ,short stature
Record Dates: First submitted 2024-04-14; First posted 2024-04-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Oral Manifestations; Short Stature
MeSH Terms: conditions — Oral Manifestations; Dwarfism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 17children with short stature
- 17 normal children

SUMMARY:
Children with short stature have been reported to show a higher prevalence of enamel hypoplasia, delayed tooth eruption, and malocclusion compared to children of normal growth status

DETAILED DESCRIPTION:
Normal growth is a process in which a single cell develops into a fully grown adult. The growth rate decelerates from the embryonic stage to adulthood, except during puberty. Most adults fall within a narrow range of stature, typically between 1.5 to 2 meters. Variations in height among children are largely determined by a set of genes inherited from their parents. These genes influence stature distribution within the normal range for nearly 95% of the population, with variation generally being benign.

Short stature in children-defined as a height-for-age below -2 standard deviations (SD) from the WHO growth reference-typically corresponding to the 2.3rd percentile, though many texts use the 3rd percentile as the cutoff. Short stature can be assessed using various anthropometric instruments. The condition may be physiological, with no abnormalities other than stature (polygenic short stature), or pathological, resulting from systemic illnesses, nutritional deficiencies, psychosocial factors, hormonal imbalances, genetic disorders, or musculoskeletal pathologies. A subset of infants born small for gestational age (SGA) may be at risk of persistent short stature.

Children with short stature have been reported to show a higher prevalence of enamel hypoplasia, delayed tooth eruption, and malocclusion compared to children of normal growth status . These oral manifestations may result from shared pathogenic mechanisms, such as nutritional deficits, systemic disturbances during enamel formation, or hormonal imbalances affecting growth and development. A clearer understanding of these associations may enhance multidisciplinary screening and care.

This study aims to investigate the prevalence and characteristics of oral manifestations in Egyptian children with short stature, contributing to the limited regional data on this topic.

ELIGIBILITY:
Inclusion Criteria:

* • - Egyptian children aged 6-12 years.
* - Diagnosed with short stature (height-for-age < -2 SD based on WHO standards).
* - Diagnosed and confirmed by a pediatric endocrinologist.

Controls:

* - Age- and sex-matched children with normal height (height-for-age between -1 and +1 SD).
* - Recruited from the same geographic and socioeconomic backgrounds.

Exclusion Criteria:

* 1- Presence of syndromic conditions (e.g., Turner syndrome, Down syndrome).
* 2- Chronic diseases (e.g., renal, cardiac, or endocrine conditions other than idiopathic short stature).
* 3- Long-term medication use known to affect growth or oral development.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged from 6 to 12 years attending National Nutrition Institute will be included in the study according to the following criteria:
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Dental enamel defects | 3 months
  using Aine's classification
Delayed dental eruption | 3 months
  using Dental eruption table
Malocclusion | 3 months
  using Angle classification
Dental caries experience | 3 months
  using def+DMF